CLINICAL TRIAL: NCT04917835
Title: Assessment of Effectiveness and Safety of Non-thermal, Atmospheric-pressure Plasma (Product Name: PLADUO) for Reduction of Sebum Excretion in Oily Facial Skin.
Brief Title: Non-thermal Plasma for Sebum Reduction in Oily Facial Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Sang Eun Lee, Assistant Professor, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-2019-0239
Record Dates: First submitted 2021-05-27; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Oily Skin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment with argon- and nitrogen-NTAPP (Experimental): PLADUO (argon- and nitrogen- non-thermal, atmospheric-pressure plasma) treatment
  Interventions: Device: PLADUO(PX1000)

INTERVENTIONS:
Device: PLADUO(PX1000) — Three sessions of argon- and nitrogen- NTAPP treatment at 1-week interval. Two passes of argon-NTAPP treatment and two passes of nitrogen-NTAPP treatment were sequentially performed in each session. Argon plasma at a pulse energy of 0.8 J/pulse with a 12 msec of pulse duration and nitrogen-plasma at a pulse energy of 0.75 J/pulse delivered with a 7 ms of pulse duration.

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of argon-and nitrogen- non-thermal, atmospheric-pressure plasma (NTAPP) for reduction of sebum excretion in healthy volunteers with oily facial skin.

DETAILED DESCRIPTION:
Excessive secretion of sebum contributes to several skin diseases associated with sebum glands, including acne. Excessive sebum secretion can damage the skin barrier function by changing the composition of skin surface lipids, leading to the abnormal keratinocyte differentiation and hyperkeratosis in the follicular ostia. Follicular hyperkeratosis can create anaerobic environment, leading to the proliferation of Propionibacterium acnes.

Recently, several energy devices targeting sebaceous glands have been developed, but there is still a need for an effective and safe therapeutic tool for hyperseborrhea. Non-thermal, atmospheric-pressure plasma (NTAPP) has various biological effects. A recent study demonstrated NTAPP-induced microscopic tissue reactions in the sebaceous glands from rat skin in vivo, suggesting that the potential effect of NTAPP on the human sebaceous gland physiology, but the relevant data are lacking. In this study, investigators aim to assess the safety and efficacy of argon- and nitrogen-NTAPP for reduction of sebum excretion in oily human facial skin.

ELIGIBILITY:
Inclusion Criteria:

1. Persons aged 19 to 40 years who are determined to have oily skin type. Skin types were classified based on the sebum measurements by using measured using a Sebumeter® (SM815; Courage+Khazaka Electronic GmbH, Cologne, Germany) according to the manufacturer's guidelines as follows: > 220 μg/cm2 on forehead and > 180 μg/cm2 on cheeks, oily type; 100-220 μg/cm2 on forehead and 70-180 μg/cm2 on cheeks, normal type; < 100 μg/cm2 on forehead and < 70 μg/cm2 on cheeks, dry type.
2. People with mild acne-like skin whose upper limit is Grade 1 (Few lesions; No nodules, papules/pustules less than 1, few comedones) and Grade 2(Mild; No nodules, papules/pustules less than 5, some comedones) of the Korean acne severity system
3. Persons who skin color of type I to III according to Fitzpatrick skin type
4. Persons who do not have inflammatory skin diseases on the facial skin
5. Persons who have heard the purpose and contents of a clinical trial and voluntarily signed the consent form prior to the clinical trial
6. Persons who can be monitored during a clinical trial period

Exclusion Criteria:

1. Persons who do not want this study or do not write a consent form
2. Persons who have a history of hypertrophic scars, keloids, etc.
3. Persons who have been using retinoid formulations within the last 1 month due to excessive sebum secretion or acne
4. Persons who have a history of receiving treatments such as lasers or fillers on your face within the last 1 month
5. Persons who is pregnant or lactating, or have a pregnancy plan within the expected trial period
6. Other cases in which the study is considered difficult due to the judgment of the principal investigator

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
Measurement of casual sebum level (μg/cm 2) | baseline, 2 weeks, 4 weeks, and 8 weeks after treatment
  The change in the casual sebum level is determined by measuring Sebumter® (SM815) from the German company Courage-khazaka. The measurement is performed in the three facial areas: forehead (mid-glabella), right and left cheeks (over the zygoma at the mid-pupillary line).
Change in the number of Ki67-and PPAR-gamma-positive sebaceous gland cells in facial tissue following treatment with argon- and nitrogen-NTAPP | baseline and 2 weeks after treatment
  Among subjects who completed the study, 2-mm skin punch biopsy specimens were obtained from zygomatic area of two volunteered subjects before and 2 weeks after argon- and nitrogen- non-thermal, atmospheric-pressure plasma treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea